CLINICAL TRIAL: NCT02621931
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing the Efficacy and Safety of 2 Dose Regimens of Subcutaneous Administration of Fremanezumab (TEV-48125) Versus Placebo for the Preventive Treatment of Chronic Migraine
Brief Title: Comparing Efficacy and Safety of 2 Dose Regimens of Subcutaneous Administration of TEV-48125 Versus Placebo for the Preventive Treatment of Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30049; 2015-004549-23 (EudraCT Number)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo
- Fremanezumab 675 mg/placebo/placebo (Experimental): Participants randomized to the fremanezumab 675 mg/placebo/placebo treatment arm received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0, and placebo as a single 1.5-mL injection on Days 28 and 56.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab 675/225/225 mg (Experimental): Participants randomized to the fremanezumab 675/225/225 mg treatment arm received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0 and 225 mg of fremanezumab as 1 active injection (225 mg/1.5 mL) on Days 28 and 56.
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab was provided as a sterile, unpreserved, aqueous solution for injection, 225 mg/1.5 mL pre-filled syringe for single-use administration. The 675 mg dose was given as 3 injections; doses of 225 mg were given as a single injection. Study drug was administered at the clinical site.
  Other Names: TEV-48125, anti-calcitonin gene-related peptide (anti-CGRP)
  Arms: Fremanezumab 675 mg/placebo/placebo; Fremanezumab 675/225/225 mg
Drug: Placebo — Placebo 1.5 mL pre-filled syringes identical in appearance to active intervention. Study drug was administered at the clinical site.
  Arms: Fremanezumab 675 mg/placebo/placebo; Placebo

SUMMARY:
The study is being conducted to evaluate two doses of TEV-48125 in adult patients with chronic migraine

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 70 years, inclusive, with migraine onset at ≤50 years of age
* Patient signs and dates the informed consent document
* Patient has history of migraine according to International Classification of Headache Disorders, or clinical judgment suggests a migraine diagnosis
* 85% e-diary compliance
* Total body weight between 99 and 250 lbs, inclusive

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Clinically significant hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, or ocular disease, at the discretion of the investigator
* Evidence or medical history of clinically significant psychiatric issues, including any suicide attempt in the past, or suicidal ideation with a specific plan in the past 2 years
* History of clinically significant cardiovascular disease or vascular ischemia (such as myocardial, neurological [eg, cerebral ischemia], peripheral extremity ischemia, or other ischemic event) or thromboembolic events (arterial or venous thrombotic or embolic events), such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism
* Known infection or history of human immunodeficiency virus, tuberculosis, or chronic hepatitis B or C infection
* Past or current history of cancer in the last 5 years, except for appropriately treated nonmelanoma skin carcinoma
* Pregnant or nursing females
* History of hypersensitivity reactions to injected proteins, including monoclonal antibodies
* Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months prior to study drug administration or 5 half-lives, whichever is longer

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (148):
- United States (94):
  - Teva Investigational Site 13628, Birmingham, Alabama
  - Teva Investigational Site 13577, Birmingham, Alabama
  - Teva Investigational Site 13606, Phoenix, Arizona
  - Teva Investigational Site 13579, Phoenix, Arizona
  - Teva Investigational Site 13602, Little Rock, Arkansas
  - Teva Investigational Site 13568, Encino, California
  - Teva Investigational Site 13546, Fullerton, California
  - Teva Investigational Site 13540, Long Beach, California
  - Teva Investigational Site 13632, Redlands, California
  - Teva Investigational Site 13571, Redondo Beach, California
  - Teva Investigational Site 13573, San Diego, California
  - Teva Investigational Site 13538, Santa Monica, California
  - Teva Investigational Site 13594, Santa Rosa, California
  - Teva Investigational Site 13595, Walnut Creek, California
  - Teva Investigational Site 13629, Aurora, Colorado
  - Teva Investigational Site 13557, Boulder, Colorado
  - Teva Investigational Site 13593, Colorado Springs, Colorado
  - Teva Investigational Site 13633, Denver, Colorado
  - Teva Investigational Site 13612, Denver, Colorado
  - Teva Investigational Site 13631, Englewood, Colorado
  - Teva Investigational Site 13563, East Hartford, Connecticut
  - Teva Investigational Site 13550, Stamford, Connecticut
  - Teva Investigational Site 13635, Bradenton, Florida
  - Teva Investigational Site 13597, Gainesville, Florida
  - Teva Investigational Site 13607, Hialeah, Florida
  - Teva Investigational Site 13559, Jacksonville, Florida
  - Teva Investigational Site 13584, Ocala, Florida
  - Teva Investigational Site 13587, Orlando, Florida
  - Teva Investigational Site 13599, Orlando, Florida
  - Teva Investigational Site 13551, Orlando, Florida
  - Teva Investigational Site 13555, Orlando, Florida
  - Teva Investigational Site 13567, Palm Beach Gardens, Florida
  - Teva Investigational Site 13553, Pembroke Pines, Florida
  - Teva Investigational Site 13616, Pinellas Park, Florida
  - Teva Investigational Site 13620, Atlanta, Georgia
  - Teva Investigational Site 13537, Atlanta, Georgia
  - Teva Investigational Site 13604, Boise, Idaho
  - Teva Investigational Site 13604, Meridian, Idaho
  - Teva Investigational Site 13585, Chicago, Illinois
  - Teva Investigational Site 13621, Chicago, Illinois
  - Teva Investigational Site 13627, Evanston, Illinois
  - Teva Investigational Site 13596, Indianapolis, Indiana
  - Teva Investigational Site 13617, Wichita, Kansas
  - Teva Investigational Site 13598, Wichita, Kansas
  - Teva Investigational Site 13566, Louisville, Kentucky
  - Teva Investigational Site 13603, Metairie, Louisiana
  - Teva Investigational Site 13582, Baltimore, Maryland
  - Teva Investigational Site 13582, Pikesville, Maryland
  - Teva Investigational Site 13590, Boston, Massachusetts
  - Teva Investigational Site 13589, New Bedford, Massachusetts
  - Teva Investigational Site 13543, Watertown, Massachusetts
  - Teva Investigational Site 13539, Ann Arbor, Michigan
  - Teva Investigational Site 13542, Golden Valley, Minnesota
  - Teva Investigational Site 13534, Kansas City, Missouri
  - Teva Investigational Site 13536, Springfield, Missouri
  - Teva Investigational Site 13619, St Louis, Missouri
  - Teva Investigational Site 13618, Fremont, Nebraska
  - Teva Investigational Site 13605, Las Vegas, Nevada
  - Teva Investigational Site 13578, Lebanon, New Hampshire
  - Teva Investigational Site 13575, Martinsville, New Jersey
  - Teva Investigational Site 13575, Raritan, New Jersey
  - Teva Investigational Site 13588, Albuquerque, New Mexico
  - Teva Investigational Site 13576, Amherst, New York
  - Teva Investigational Site 13565, Plainview, New York
  - Teva Investigational Site 13544, Greensboro, North Carolina
  - Teva Investigational Site 13574, Greensboro, North Carolina
  - Teva Investigational Site 13545, Raleigh, North Carolina
  - Teva Investigational Site 13609, Akron, Ohio
  - Teva Investigational Site 13634, Akron, Ohio
  - Teva Investigational Site 13533, Cincinnati, Ohio
  - Teva Investigational Site 13624, Cincinnati, Ohio
  - Teva Investigational Site 13569, Cleveland, Ohio
  - Teva Investigational Site 13626, Columbus, Ohio
  - Teva Investigational Site 13625, Mogadore, Ohio
  - Teva Investigational Site 13561, Oklahoma City, Oklahoma
  - Teva Investigational Site 13601, Eugene, Oregon
  - Teva Investigational Site 13591, Jenkintown, Pennsylvania
  - Teva Investigational Site 13554, Philadelphia, Pennsylvania
  - Teva Investigational Site 13608, Uniontown, Pennsylvania
  - Teva Investigational Site 13615, Greer, South Carolina
  - Teva Investigational Site 13556, Mt. Pleasant, South Carolina
  - Teva Investigational Site 13560, Bristol, Tennessee
  - Teva Investigational Site 13532, Nashville, Tennessee
  - Teva Investigational Site 13552, Nashville, Tennessee
  - Teva Investigational Site 13541, Austin, Texas
  - Teva Investigational Site 13623, Dallas, Texas
  - Teva Investigational Site 13611, Plano, Texas
  - Teva Investigational Site 13572, San Antonio, Texas
  - Teva Investigational Site 13614, Murray, Utah
  - Teva Investigational Site 13581, West Jordan, Utah
  - Teva Investigational Site 13630, Virginia Beach, Virginia
  - Teva Investigational Site 13564, Seattle, Washington
  - Teva Investigational Site 13586, Seattle, Washington
  - Teva Investigational Site 13600, Morgantown, West Virginia
- Canada (5):
  - Teva Investigational Site 11124, Hamilton, Ontario
  - Teva Investigational Site 11120, Calgary
  - Teva Investigational Site 11121, Montreal
  - Teva Investigational Site 11122, Newmarket
  - Teva Investigational Site 11123, Sarnia
- Czechia (6):
  - Teva Investigational Site 54144, Brno
  - Teva Investigational Site 54141, Kunratice
  - Teva Investigational Site 54145, Pardubice
  - Teva Investigational Site 54143, Prague
  - Teva Investigational Site 54146, Prague
  - Teva Investigational Site 54142, Prague
- Finland (3):
  - Teva Investigational Site 40018, Helsinki
  - Teva Investigational Site 40017, Helsinki
  - Teva Investigational Site 40016, Turku
- Israel (6):
  - Teva Investigational Site 80096, Holon
  - Teva Investigational Site 80099, Jerusalem
  - Teva Investigational Site 80098, Nahariya
  - Teva Investigational Site 80097, Netanya
  - Teva Investigational Site 80100, Ramat Gan
  - Teva Investigational Site 80095, Tel Aviv
- Japan (18):
  - Teva Investigational Site 84072, Chofu-shi
  - Teva Investigational Site 84064, Chofu-shi
  - Teva Investigational Site 84066, Kagoshima
  - Teva Investigational Site 84069, Kai
  - Teva Investigational Site 84069, Kaisho
  - Teva Investigational Site 84073, Kawasaki
  - Teva Investigational Site 84073, Kawasaki-shi
  - Teva Investigational Site 84067, Kyoto
  - Teva Investigational Site 84062, Osaka
  - Teva Investigational Site 84070, Saitama
  - Teva Investigational Site 84070, Saitama-shi
  - Teva Investigational Site 84061, Sendai
  - Teva Investigational Site 84065, Shimotsuma
  - Teva Investigational Site 84068, Shizuoka
  - Teva Investigational Site 84065, Tochigi
  - Teva Investigational Site 84064, Tokyo
  - Teva Investigational Site 84071, Toyonaka
  - Teva Investigational Site 84071, Toyonaka-shi
- Poland (5):
  - Teva Investigational Site 53364, Krakow
  - Teva Investigational Site 53363, Krakow
  - Teva Investigational Site 53366, Lublin
  - Teva Investigational Site 53365, Poznan
  - Teva Investigational Site 53367, Warsaw
- Russia (7):
  - Teva Investigational Site 50399, Kazan'
  - Teva Investigational Site 50395, Kazan'
  - Teva Investigational Site 50394, Moscow
  - Teva Investigational Site 50400, Moscow
  - Teva Investigational Site 50398, Nizhny Novgorod
  - Teva Investigational Site 50396, Nizhny Novgorod
  - Teva Investigational Site 50397, Ufa
- Spain (4):
  - Teva Investigational Site 31207, Madrid
  - Teva Investigational Site 31208, Pamplona
  - Teva Investigational Site 31205, Valladolid
  - Teva Investigational Site 31206, Zaragoza

REFERENCES:
- [Derived] McAllister P, Cohen JM, Campos VR, Ning X, Janka L, Barash S. Impact of fremanezumab on disability outcomes in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. J Headache Pain. 2022 Aug 29;23(1):112. doi: 10.1186/s10194-022-01438-4. PMID 36038833
- [Derived] Diener HC, McAllister P, Jurgens TP, Kessler Y, Ning X, Cohen JM, Campos VR, Barash S, Silberstein SD. Safety and tolerability of fremanezumab in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. Cephalalgia. 2022 Jul;42(8):769-780. doi: 10.1177/03331024221076485. Epub 2022 Mar 25. PMID 35331009
- [Derived] Nahas SJ, Naegel S, Cohen JM, Ning X, Janka L, Campos VR, Krasenbaum LJ, Holle-Lee D, Kudrow D, Lampl C. Efficacy and safety of fremanezumab in clinical trial participants aged >/=60 years with episodic or chronic migraine: pooled results from 3 randomized, double-blind, placebo-controlled phase 3 studies. J Headache Pain. 2021 Nov 24;22(1):141. doi: 10.1186/s10194-021-01351-2. PMID 34819017
- [Derived] Silberstein SD, Cohen JM, Yang R, Gandhi SK, Du E, Jann AE, Marmura MJ. Treatment benefit among migraine patients taking fremanezumab: results from a post hoc responder analysis of two placebo-controlled trials. J Headache Pain. 2021 Jan 7;22(1):2. doi: 10.1186/s10194-020-01212-4. PMID 33413075
- [Derived] Silberstein SD, Cohen JM, Seminerio MJ, Yang R, Ashina S, Katsarava Z. The impact of fremanezumab on medication overuse in patients with chronic migraine: subgroup analysis of the HALO CM study. J Headache Pain. 2020 Sep 21;21(1):114. doi: 10.1186/s10194-020-01173-8. PMID 32958075
- [Derived] Lipton RB, Cohen JM, Gandhi SK, Yang R, Yeung PP, Buse DC. Effect of fremanezumab on quality of life and productivity in patients with chronic migraine. Neurology. 2020 Aug 18;95(7):e878-e888. doi: 10.1212/WNL.0000000000010000. Epub 2020 Aug 3. PMID 32747522
- [Derived] Winner PK, Spierings ELH, Yeung PP, Aycardi E, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y. Early Onset of Efficacy With Fremanezumab for the Preventive Treatment of Chronic Migraine. Headache. 2019 Nov;59(10):1743-1752. doi: 10.1111/head.13654. Epub 2019 Nov 1. PMID 31675102
- [Derived] Silberstein SD, Dodick DW, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Fremanezumab for the Preventive Treatment of Chronic Migraine. N Engl J Med. 2017 Nov 30;377(22):2113-2122. doi: 10.1056/NEJMoa1709038. PMID 29171818

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3148 patients with migraine provided written informed consent and were screened for entry into either Study TV48125-CNS-30049 or Study TV48125-CNS-30050. Of the 3148 screened, 1130 met entry criteria, including criteria for chronic migraine and diary compliance during the run-in period, and were randomized into this study.
Groups:
- Placebo: Participants randomized to the placebo treatment arm received three 1.5-mL placebo injections at Day 0 and a single 1.5-mL placebo injection at Days 28 and 56 .
Period: Overall Study
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Started | 375 | 376 | 379
Safety and ITT Populations | 375 | 376 | 379
Full Analysis Set | 371 | 375 | 375
Completed | 342 | 349 | 343
Not Completed | 33 | 27 | 36
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 8 | 5 | 7
Not completed — Withdrawal by Subject | 12 | 10 | 11
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Noncompliance to study procedures | 0 | 1 | 2
Not completed — Lost to Follow-up | 8 | 7 | 10
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Other | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg | Total
Number analyzed (Participants) | 375 | 376 | 379 | 1130
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.03) | 42.0 (12.37) | 40.6 (11.95) | 41.3 (12.12)
Age, Customized [Count of Participants; unit: Participants]
  18-45 years | 229 | 218 | 248 | 695
  46-65 years | 143 | 149 | 123 | 415
  >65 years | 3 | 9 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 331 | 330 | 991
  Male | 45 | 45 | 49 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 303 | 293 | 297 | 893
  Black | 29 | 33 | 37 | 99
  Asian | 40 | 40 | 41 | 121
  American Indian or Alaska Native | 0 | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Other | 2 | 4 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not HIspanic or Latino | 343 | 352 | 338 | 1033
  Hispanic or Latino | 32 | 22 | 41 | 95
  Unknown | 0 | 1 | 0 | 1
  Not reported | 0 | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] — Population: Two participants were missing baseline weight data
  kg
    number analyzed (Participants) | 375 | 376 | 377 | 1128
    (all) | 72.6 (15.58) | 72.4 (15.79) | 72.5 (16.36) | 72.5 (15.90)
Time Since Initial Migraine Diagnosis [Mean (Standard Deviation); unit: years] | 19.9 (12.86) | 19.7 (12.84) | 20.1 (11.98) | 19.9 (12.55)
Preventative Medication Use During Baseline Period [Count of Participants; unit: Participants] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. During randomization, patients were stratified based on sex, country, and baseline preventive migraine medication use (yes, no) to ensure balance for the covariates.
  Participants
    Yes | 77 | 77 | 85 | 239
    No | 298 | 299 | 294 | 891
Total Number of Headache Days of Any Duration And Any Severity During the 28 Day Baseline Period [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device.
  days | 20.3 (4.19) | 20.4 (3.93) | 20.3 (4.26) | 20.3 (4.13)
Number of Headache Days of At Least Moderate Severity [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. Headache severity was subjectively rated by the patient as mild, moderate or severe.
  days | 13.3 (5.82) | 13.2 (5.47) | 12.8 (5.80) | 13.1 (5.70)
Number of Migraine Days [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. Migraine headaches are as defined in The International Classification of Headache Disorders 3rd edition (ICHD-3).
  days | 16.4 (5.15) | 16.2 (4.88) | 16.0 (5.19) | 16.2 (5.97)
Number of Days of Use of Any Acute Headache Medications [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information (including information about use of headache medications) was captured daily throughout study participation using the electronic headache diary device.
  days | 13.0 (6.92) | 13.1 (6.79) | 13.1 (7.20) | 13.1 (6.96)
Headache Impact Test (HIT-6) Disability Score [Mean (Standard Deviation); unit: units on a scale] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. HIT-6 measures the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning, and psychological distress. It also assesses headache severity. Scores range from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the patient. Scores ≥60 indicate severe impact. Population: HIT-6 was not assessed at baseline for some patients.
  units on a scale
    number analyzed (Participants) | 373 | 370 | 377 | 1120
    (all) | 64.1 (4.80) | 64.3 (4.74) | 64.6 (4.42) | 64.3 (4.65)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Average Number of Headache Days of At Least Moderate Severity During the 12-Week Period After the First Dose of Study Drug
Description: Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) where the patient (using the electronic headache diary device) reports: - a day with headache pain that lasts ≥4 hours with a peak severity of at least moderate severity or - a day when the patient used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as post-baseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set (FAS) included those in the intent to treat (ITT) population who received at least 1 dose of study drug and had at least 10 days of post-baseline efficacy assessments on the primary endpoint.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 371 | 375 | 375
days | -2.5 [-5.6 to 0.0] | -4.2 [-7.7 to -1.7] | -4.5 [-7.8 to -1.7]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Due to the deviation from the normal distribution assumption of the data, the primary analysis was conducted using the Wilcoxon rank-sum test as outlined in the statistical analysis plan (SAP); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance; LSM difference from placebo = -1.8, 95% CI 2-sided [-2.46 to -1.15], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Due to the deviation from the normal distribution assumption of the data, the primary analysis was conducted using the Wilcoxon rank-sum test as outlined in the SAP; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance; LSM difference from placebo = -2.1, 95% CI 2-sided [-2.76 to -1.45], Standard Error of Mean 0.33

2. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents usual activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 375 | 376 | 379
Participants
  Any TEAE | 240 | 265 | 270
  Severe TEAE | 20 | 14 | 15
  Treatment-related TEAE | 159 | 186 | 194
  Serious TEAE | 6 | 3 | 5
  Death | 0 | 1 | 0
  TEAE leading to discontinuation | 8 | 5 | 7

3. Secondary Outcome: Change From Baseline in the Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Study Drug
Description: A migraine day was defined as when at least 1 of the following situations occurred: - a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for migraine with or without aura - a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing - a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as post-baseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: migraine days / month
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 371 | 375 | 375
migraine days / month | -3.2 (0.35) | -4.9 (0.35) | -5.0 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Test type: Superiority; p < 0.0001, ANCOVA — 0.05 level of significance; LSM difference from placebo = -1.7, 95% CI 2-sided [-2.48 to -0.97], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Test type: Superiority; p < 0.0001, ANCOVA — 0.05 level of significance; LSM difference from placebo = -1.8, 95% CI 2-sided [-2.61 to -1.09], Standard Error of Mean 0.39

4. Secondary Outcome: Percentage of Participants With At Least 50% Reduction In Monthly Average Number of Headache Days of At Least Moderate Severity
Description: Responder rates were defined as the percentage of total subjects who reached at least a 50% reduction in the monthly average of headache days (as subjectively reported by participants in the study diary) of at least moderate severity relative to the baseline period. For the overall analysis (Month 1-3), patients who discontinued early were considered non-responders. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The percentage reduction in monthly average is calculated as: ((baseline value - post-baseline value) / baseline value) * 100.
Time Frame: Baseline (Days -28 to Day -1), Treatment: Month 1, Month 2, Month 3, Month 1-3 (Days 1 - Week 12)
Population: FAS. One participant in the Placebo and Fremanezumab 675/225/225 mg treatment arms had 0 headache days of >= moderate severity during baseline and treatment and therefore was not included.
Measure: Number; unit: percentage of total participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 370 | 375 | 374
percentage of total participants
  Month 1 | 21.6 | 41.3 | 40.0
  Month 2: number analyzed (Participants) | 355 | 365 | 361
  Month 2 | 24.3 | 39.7 | 41.9
  Month 3: number analyzed (Participants) | 342 | 350 | 345
  Month 3 | 26.4 | 40.5 | 44.5
  Overall - Months 1-3 | 18.1 | 37.6 | 40.8
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 1: Active 675/placebo/placebo to Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — 0.05 level of significance. P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Month 1: Active 675/225/225 to Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Month 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 3; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Month 3; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Overall; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Overall; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in the Monthly Average Number of Days of Use of Any Acute Headache Medicine During the 12 Week Period After the First Dose of Study Drug
Description: Participants recorded any migraine medications (name of drug, number of tablets/capsules, and the dose in milligrams per tablet/capsule) taken on each day in their electronic headache diary device. Acute migraine-specific medication included triptans or ergots. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as post-baseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Placebo: Participants randomized to the placebo treatment arm received three 1.5-mL placebo injections at Day 0 and a single 1.5-mL placebo injection at Days 28 and 56.
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 371 | 375 | 375
days | -2.0 [-5.3 to 0.2] | -3.6 [-7.3 to -0.7] | -4.2 [-7.6 to -1.1]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

6. Secondary Outcome: Change From Baseline in the Number of Headache Days of At Least Moderate Severity During the 4 Week Period After the First Dose of Study Drug
Description: Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) where the patient (using the electronic headache diary device) reports: - a day with headache pain that lasts ≥4 hours with a peak severity of at least moderate severity or - a day when the patient used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration. The change is calculated as post-baseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 4)
Population: Full analysis set (FAS) included those in the ITT population who received at least 1 dose of study drug and had at least 10 days of post-baseline efficacy assessments on the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: days
Groups:
- Fremanezumab 675 mg: Participants randomized to both fremanezumab treatment arms received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0. Later treatments are beyond the timeframe for this outcome. Therefore the data from both active treatment arms were combined for this comparison.
Arm/Group | Placebo | Fremanezumab 675 mg
Number analyzed (Participants) | 371 | 750
days | -2.3 (0.33) | -4.6 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg; Test type: Superiority; p < 0.0001, ANCOVA — 0.05 level of significance; LSM difference from placebo = -2.3, 95% CI 2-sided [-2.95 to -1.73], Standard Error of Mean 0.31

7. Secondary Outcome: Change From Baseline in the Monthly Average Number of Headache Days of At Least Moderate Severity During the 12 Week Period After the First Dose of Study Medication in Patients Not Receiving Concomitant Preventive Migraine Medications
Description: A subset of patients (specified in the protocol not to exceed 30%) were allowed to use 1 concomitant migraine preventive medication. This outcome only includes those participants who did not take concomitant preventive migraine medication during this study. Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of >= moderate severity was defined as a calendar day where the patient (using the electronic headache diary device) reports: - a day with headache pain that lasts ≥4 hours with a peak severity of >= moderate severity or - a day when the patient used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. Change is post-baseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: FAS of participants who did not receive concomitant preventive migraine medications.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 294 | 298 | 290
days | -2.4 [-5.3 to 0.0] | -4.4 [-8.0 to -1.7] | -4.6 [-7.8 to -1.5]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

8. Secondary Outcome: Change From Baseline in Migraine-Related Disability Score, As Measured by the 6-Item Headache Impact Test (HIT) At Week 12
Description: The HIT-6 was developed by Kosinski et al (2003) as a short form for reliably assessing the adverse headache impact in clinical practice and clinical research settings. The questionnaire measures the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning, and psychological distress. It also assesses headache severity. Scores range from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the patient, i.e. scores ≤49 represent little or no impact, scores between 50 and 55 represent some impact, scores between 56 and 59 represent substantial impact; and scores ≥60 indicate severe impact. Negative change from baseline values indicate less adverse impact of headache.
Time Frame: Baseline, 12 weeks
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 371 | 375 | 375
units on a scale | -4.0 [-7.0 to 0.0] | -5.0 [-10.0 to -2.0] | -6.0 [-11.0 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 675/225/225 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

9. Secondary Outcome: Electrocardiogram (ECG) Findings Shifts From Baseline to Overall
Description: 12-lead ECGs were performed before other assessments (eg, blood draws and administration of questionnaires) and performed in triplicate. The worst post-baseline finding for the participant is summarized. Only participants with both baseline and post-baseline ECGs are included. The ECG was evaluated by the investigator at the time of recording (signed and dated), and the printout was kept in the source documentation file. When potentially clinically significant findings were detected by the investigator, a cardiologist at a central diagnostic center was consulted for a definitive interpretation. Any ECG finding that was judged by the investigator as a potentially clinically significant change (worsening) compared with a baseline value was considered an adverse event. - NCS = abnormal, not clinically significant. - CS= abnormal, clinically significant. Shift format is: baseline finding / worst post-baseline finding.
Time Frame: Baseline (Day 0), Treatment Week 12 (or endpoint)
Population: Safety population of participants with both baseline and post-treatment ECGs.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 360 | 361 | 362
Participants
  Normal / Normal | 215 | 220 | 223
  Normal / NCS | 54 | 48 | 43
  Normal / CS | 1 | 0 | 0
  NCS / Normal | 31 | 34 | 34
  NCS / NCS | 59 | 59 | 62
  NCS / CS | 0 | 0 | 0
  CS / Normal | 0 | 0 | 0
  CS / NCS | 0 | 0 | 0
  CS / CS | 0 | 0 | 0

10. Secondary Outcome: Participants With Vital Signs Potentially Clinically Significant Abnormal Values
Description: Vital signs were performed before other assessments (eg, blood draws and administration of questionnaires). Vital signs with potentially clinically significant abnormal findings included: - Pulse Rate High: >=120 and increase of >=15 beats per minute - Pulse Rate Low: <=50 and decrease of >=15 beats per minute - Systolic Blood Pressure Low: <=90 mmHg and decrease of >=20 mmHg - Diastolic Blood Pressure High: >=105 mmHg and increase of >=15 mmHg - Diastolic Blood Pressure Low: <=50 mmHg and decrease of >=15 mmHg - Respiratory Rate Low: <10 breaths / minute
Time Frame: Treatment Days 28, 56 and 84 (or endpoint). Changes from previous reading may reflect the baseline reading performed on Day 0.
Population: Safety population of participants with both baseline and post-treatment values for each vital sign.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 366 | 373 | 372
Participants
  Participants with at least 1 abnormality | 7 | 10 | 14
  Pulse Rate High | 0 | 0 | 1
  Pulse Rate Low | 1 | 1 | 0
  Systolic Blood Pressure Low | 2 | 4 | 6
  Diastolic Blood Pressure High | 1 | 2 | 3
  Diastolic Blood Pressure Low | 0 | 1 | 2
  Respiratory Rate Low | 3 | 2 | 3

11. Secondary Outcome: Participants With Serum Chemistry and Hematology Potentially Clinically Significant Abnormal Results
Description: Serum chemistry and hematology laboratory tests with potentially clinically significant abnormal findings included: - Blood Urea Nitrogen (BUN) High: >=10.71 mmol/L - Creatinine High: >=177 umol/L - Bilirubin High: >=34.2 umol/L - Alanine Aminotransferase (ALT): >=3*upper limit of normal (ULN) - Aspartate Aminotransferase (AST): >=3*upper limit of normal (ULN) - Gamma Glutamyl Transferase (GGT): >=3*upper limit of normal (ULN) - Hemoglobin: Male: <115 g/L or Female: <=95 g/L - Hematocrit: Male: <0.37 L/L or Female: <0.32 L/L - Leukocytes: >=20*10^9/L or <=3*10^9/L - Eosinophils/Leukocytes: >=10% - Platelets: >=700*10^9/L or <=75*10^9/L
Time Frame: Treatment Days 28, 56 and 84 (or endpoint)
Population: Safety population of participants with at least one post-baseline result for the tests
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 366 | 373 | 371
Participants
  BUN | 1 | 1 | 1
  Creatinine | 2 | 0 | 0
  Bilirubin | 0 | 2 | 0
  ALT | 2 | 2 | 7
  AST | 0 | 3 | 4
  GGT | 7 | 7 | 8
  Hemoglobin | 2 | 5 | 3
  Hematocrit | 8 | 9 | 7
  Leukocytes | 2 | 9 | 5
  Eosinophils/Leukocytes | 4 | 5 | 4
  Platelets: number analyzed (Participants) | 366 | 371 | 371
  Platelets | 1 | 2 | 0

12. Secondary Outcome: Participants With Urinalysis Laboratory Tests Potentially Clinically Significant Abnormal Results
Description: Urinalysis with potentially clinically significant abnormal findings included: - Blood: >=2 unit increase from baseline - Urine Glucose (mg/dL): >=2 unit increase from baseline - Ketones (mg/dL): >=2 unit increase from baseline - Urine Protein (mg/dL): >=2 unit increase from baseline
Time Frame: Treatment Days 28, 56 and 84 (or endpoint). Changes from previous reading reflect the baseline reading performed on Day 0.
Population: Safety population of participants with at least one post-baseline result for the tests.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 365 | 373 | 372
Participants
  Participants with at least 1 abnormality | 78 | 57 | 68
  Blood | 33 | 32 | 35
  Urine glucose | 7 | 7 | 5
  Ketones | 7 | 7 | 7
  Urine protein | 40 | 19 | 34

13. Secondary Outcome: Prothrombin Time Shifts From Baseline to Endpoint
Description: Shifts in prothrombin time from baseline to endpoint were summarized using patient counts grouped into three categories: - Low (below normal range) - Normal (within the normal range of 9.4 to 12.5 seconds) - High (above normal range) Shift format is: baseline finding / endpoint finding
Time Frame: Baseline (Day 0), Treatment Endpoint (Week 12)
Population: Safety population of participants with both baseline and post-treatment values
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 366 | 373 | 370
Participants
  Low / Low | 0 | 0 | 0
  Low / Normal | 2 | 0 | 1
  Low / High | 0 | 0 | 0
  Normal / Low | 0 | 1 | 2
  Normal / Normal | 330 | 318 | 327
  Normal / High | 13 | 17 | 19
  High / Low | 0 | 0 | 0
  High / Normal | 14 | 19 | 12
  High / High | 7 | 18 | 9

14. Secondary Outcome: Injection Site Reaction Adverse Events
Description: Counts of participants who reported treatment-emergent injection site reactions as AEs are summarized. Preferred terms from MedDRA version 18.1 are offered without a threshold applied.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 375 | 376 | 379
Participants
  Participants with >= 1 injection site reaction | 151 | 176 | 183
  Injection site pain | 104 | 114 | 99
  Injection site induration | 68 | 74 | 90
  Injection site erythema | 60 | 80 | 75
  Injection site haemorrhage | 10 | 7 | 8
  Injection site pruritus | 0 | 6 | 8
  Injection site rash | 0 | 4 | 3
  Injection site bruising | 2 | 1 | 2
  Injection site swelling | 0 | 2 | 1
  Injection site dermatitis | 0 | 1 | 0
  Injection site discomfort | 0 | 1 | 0
  Injection site haematoma | 0 | 0 | 1
  Injection site hypoaesthesia | 0 | 0 | 1
  Injection site inflammation | 0 | 0 | 1
  Injection site oedema | 0 | 1 | 0
  Injection site paraesthesia | 0 | 0 | 1
  Injection site urticaria | 2 | 0 | 1
  Injection site warmth | 2 | 0 | 1

15. Secondary Outcome: Participants With Positive Electronic Columbia Suicide Severity Rating Scale (eC-SSRS) Results After the First Dose of Study Drug
Description: The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) was used to assess the participant's suicidal ideation (severity and intensity) and behavior (Posner et al 2011). Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
  The eC-SSRS Baseline/Screening version was completed by the participant at baseline, and the eC-SSRS Since Last Visit version was completed by the participant at all other time points. Any positive findings on the eC-SSRS Since Last Visit version required evaluation by a physician or doctoral-level psychologist. Findings after the first dose of study drug using the eC-SSRS Since Last Visit version are summarized.
Time Frame: Baseline (Day 0), Treatment Days 28, 56, 84
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
Number analyzed (Participants) | 375 | 376 | 379
Participants
  Participants with positive eC-SSRS responses | 1 | 1 | 1
  Specific finding: interrupted suicide attempt | 1 | 1 | 0
  Specific finding: suicidal ideation | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Groups:
- Placebo: Participants randomized to receive placebo received three 1.5-mL placebo injections at Day 0 and a single 1.5-mL placebo injection at Days 28 and 56.
- Fremanezumab 675 mg/Placebo/Placebo: Participants randomized to receive fremanezumab 675 mg/placebo/placebo received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0, and placebo as a single 1.5-mL injection on Days 28 and 56.
- Fremanezumab 675/225/225 mg: Participants randomized to receive fremanezumab 675/225/225 mg received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0 and 225 mg of fremanezumab as 1 active injection (225 mg/1.5 mL) on Days 28 and 56.
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 675/225/225 mg
All-Cause Mortality (participants affected / at risk) | 0/375 | 1/376 | 0/379
Serious Adverse Events (participants affected / at risk) | 6/375 | 3/376 | 5/379
Other Adverse Events (participants affected / at risk) | 160/375 | 185/376 | 178/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=375) | Fremanezumab 675 mg/Placebo/Placebo (N=376) | Fremanezumab 675/225/225 mg (N=379)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=375) | Fremanezumab 675 mg/Placebo/Placebo (N=376) | Fremanezumab 675/225/225 mg (N=379)
Injection site erythema (General disorders) | 60 (129) | 80 (172) | 75 (166)
Injection site induration (General disorders) | 68 (130) | 74 (159) | 90 (196)
Injection site pain (General disorders) | 104 (288) | 114 (296) | 99 (271)
Nasopharyngitis (Infections and infestations) | 20 (24) | 19 (20) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02621931/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT02621931/SAP_001.pdf